CLINICAL TRIAL: NCT02597205
Title: TAKEmeds Program: The Adherence and Knowledge Exchange Heart and Stroke Medicines Study
Brief Title: The Adherence and Knowledge Exchange Heart and Stroke Medicines Study
Acronym: TAKEmeds
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Duke Kunshan University (Other)
Collaborators: Population Health Research Institute (Other); Fudan University (Other); Hainan Provincial Nongken General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014HHSC0016
Record Dates: First submitted 2015-06-19; First posted 2015-11-05 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Myocardial Infarction
Keywords: Medical adherence; Lifestyle modification; Mobile Health; Secondary Prevention
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mobile app (Experimental): Multi-faceted intervention for physicians and patients respectively: physician-facing app and patient-facing messages
  Interventions: Behavioral: physician-facing app and patient-facing messages

INTERVENTIONS:
Behavioral: physician-facing app and patient-facing messages — A physician-facing app was designed to help physicians with recruiting and managing patients and with evidence-based medications prescription. Messages were also developed to send to patients to improve their medical adherence and modify lifestyle.

SUMMARY:
The overarching goal of this program to increase the use of evidence-based, secondary-prevention medications and promote healthy lifestyles among myocardial infarction (MI) patients through using provider-facing mobile app and patients-facing text messages.

DETAILED DESCRIPTION:
Background:

Cardiovascular disease (CVD) affects half of all individuals over their lifetime.CVD is the leading cause of all non-communicable disease (NCD) deaths, and is projected to increase by 15% worldwide between 2010 and 2020. A wealth of evidence and international guidelines support the use of low-cost, evidence-based medication, for the management of established CVD.

Study aim:

1. To develop and test the usability of a multifaceted, information-technology intervention among patients with a history of myocardial infarction (MI) and their healthcare providers.
2. To develop, contextualize and assess the efficacy of patient-directed text messages as a means of improving medication adherence among myocardial Infraction patients in Shanghai, China.
3. To test the usability and efficacy of text message reminders aimed at modifying major health risk behaviors including smoking and diet among MI patients.

Methods:

Study design overview:

This is a short-term, quasi-experimental, pre-post intervention study designed to evaluate the feasibility and effectiveness of using mobile phone app and text messaging as a means to improve adherence to medication for secondary prevention, promote behavior change, and reduce risk factors among MI patients.

Study setting and study team:

The study is going to be conducted in Shanghai and Haikou, Hainan, China. There are four academic collaborating institutions in this study: Global Health Research Center, Duke Kunshan University (DKU), China, Population Health Research Institution (PHRI), Canada and School of Public Health, Fudan University, China and Hainan Nongken General Hospital, China.

The DKU research team plays the leading role to design the study, develop the app and messages and oversee the entire implementation process. The PHRI research team will primarily work with the DKU research team on the physician-facing app and patient-facing messages development. The Fudan and Hainan research team will be responsible for local implementation.

Pre-intervention preparation:

Development of provider software application: To understand the actual needs and barriers that physicians face in using the app, the DKU research team will conduct assessment among physicians in the three community healthcare centers. The assessment is done through a short survey and key informant interview. Information from the survey and interviews will inform app design and development decisions.

Development of patient-centered message bank: The DKU research team will work with the PHRI research team to develop the message bank through literature review search. The message bank will cover five domains to help MI patients with medical adherence and lifestyle modification: 1) medical adherence; 2) diet; 3) exercise; 4) smoking cessation; 5) general heart health (see appendix 4 for the messages). To contextualize the messages and ensure its comprehensibility to patients, the Fudan and Hainan research team will invite physicians to validate the message (see appendix 5 for the message validation survey). Physicians will be asked to score each message in terms of its likability and comprehensibility. Two messages in each domain with the lowest score will be deleted. Considering that reading texts might be difficult for some patients, voice message option is also available for patients to choose. The contents of both the texts and voice messages are identical.

Intervention:

The study is designed to have two interventions targeting physicians and patients respectively. Only one community healthcare center will receive the intervention and the intervention period is designed to be 12 weeks. The Fudan and Hainan research team will be responsible for recruiting physicians and each physician will recruit MI patients to participate in the study. Physicians play dual role in this study: 1) as subjects who will use the app to prescribe medications and 2) as collaborators who will help recruit patients and collect their baseline data. The DKU research team will train the physicians how to use the app before they start to recruit patients.

1. Provider-level intervention:

   Physicians will use the smart phone application, specifically designed for this study, to help them with medications prescription and patient recruitment. The prescription recommendations are based on the NICE (National Institute for Health and Care Excellence) guidelines 2014 in MI secondary prevention.
2. Patient-level intervention:

Patients that are eligible to participate will receive automated, periodic evidence-based text messages about consistent medication use and lifestyle modification via text-messaging. They will receive standard ongoing care as well as regular unidirectional text messages via text or voice message over a 12 week period.

Process Evaluation:

Qualitative research methods will be used to obtain feedback from both the providers and the patients on the physician app and the short messaging system (SMS). To assess whether the intervention is implemented as planned and to gain their user feedback, the DKU, Fudan and Hainan research team will conduct phone and face-to-face interviews respectively in the middle and at the end of the intervention. All questions will be open-ended allowing participants to raise important issues even if they are not covered in our original topic guide. Four physicians and eight patients (two from each physician) will be invited to participate in the process evaluation interview. The mid-term evaluation (between 4-6 weeks after the intervention begins) are all one-on-one in-depth interviews. The final-term evaluation will consist of one focus group discussion among the four physicians and individual interviews to patients.

Data management and analysis:

Questionnaires require translation before coding and further data analysis can occur. In addition to coding and translation, interviews and focus groups will both be recorded and require transcription. All data entry will be performed by the Fudan and Hainan research team and will occur as close to the time of data collection to ensure accuracy.

Descriptive analysis will be used to describe the rate of adherence among the patients. Percentage differences in the proportion of patients who adhered to medication use and those who did not adhere to the medication use will be compared. Characteristics will be compared at baseline and after follow-up by using independent t tests for continuous variables (physical activity and diet) or chi-square tests for categorical variables (smoking status). Analyses will be performed using stata, version 12. Lastly, the interview and focus groups transcriptions will be coded for emerging themes using QSR Nvivo.

Risks and benefits:

This study offers participants the prospect of direct benefits: 1) it may potentially improve patient medical adherence; 2) it may potentially help patients build healthy lifestyle; 3) it may give guidance for physicians on evidence-based medicines prescription; 4) it may facilitate interactions between patients and physicians.

No foreseeable risks are anticipated for physicians. As for patients, one concern is that the exercise promotion messages, if taken without cautions, may to some degree increase the risk of heart attack for some patients. To eliminate this concern, the text messages suggest patients consult their doctors first before taking any exercise to reduce such risk to minimal. The risk of possible breach of confidentiality is addressed through using vigorous methods to protect the identity of subjects. After the data are collected, entered, and digitized, the investigators will store identifiable information in a separate data set and remove all such information from the main database (same to the information collected at the pre-intervention stage). The app will generate a unique identification number (ID) for each physician and patient for confidentiality use. Linkage will be through the study ID and performed only when necessary. Baseline and follow-up surveys will be linked by study ID only. As for the information collected on the app, they cannot be accessed without entering the password set by the physicians themselves. Only physicians, programmers and DKU research team members have access to it when necessary.

ELIGIBILITY:
Inclusion Criteria:

* Physicians who: 1) manage MI patients; 2) are interested in and consent to participate in this project; 3) have an Android-based smart phone;
* Patients who: 1) if they have suffered from a myocardial infraction; 2) they are physical and mentally able to manage their MI conditions; 3) they own a mobile telephone with the ability to read text messages or receive voice messages, and 4) willing to provide informed consent.

Exclusion Criteria:

* Physicians who i) do not have an Android smart phone or not being able to use one; ii) do not managing MI patients; iii) current participating in another study.
* Patients who are: 1) not being able to use a cellphone; 2) severally ill; 3) current participating in another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Medical adherence change | Three months
  Score change measured by the well-validated 4-item Morisky Green Levine Scale

SECONDARY OUTCOMES:
Change in diet | Three months
  Measured by the BRFSS: Fruit and Vegetable Module
Change in exercise | Three months
  Measured by the International Physical Activity Questionnaire
Change in smoking habit | Three months
  Measured by the Tobacco Questions for Surveys, World Health Organization

CONTACTS AND LOCATIONS:
Overall Officials: JD Schwalm, MD, Principal Investigator — Population Health Research Institute, Hamilton Health Sciences Corporation, Canada
Locations (2):
- China (2):
  - Hainan Nongken General Hospital, Haikou, Hainan
  - Shanghai Xietu Street Community Healthcare Center, Shanghai, Shanghai Municipality

REFERENCES:
- [Background] Selected leading causes of death.: Statistics Canada; 2005.
- [Background] Global Status Report on Non-Communicable Diseases 2010. Geneva World Health Organization; 2011.
- [Background] Lloyd-Jones DM, Leip EP, Larson MG, D'Agostino RB, Beiser A, Wilson PW, Wolf PA, Levy D. Prediction of lifetime risk for cardiovascular disease by risk factor burden at 50 years of age. Circulation. 2006 Feb 14;113(6):791-8. doi: 10.1161/CIRCULATIONAHA.105.548206. Epub 2006 Feb 6. PMID 16461820
- [Background] Alwan A, Maclean DR, Riley LM, d'Espaignet ET, Mathers CD, Stevens GA, Bettcher D. Monitoring and surveillance of chronic non-communicable diseases: progress and capacity in high-burden countries. Lancet. 2010 Nov 27;376(9755):1861-8. doi: 10.1016/S0140-6736(10)61853-3. Epub 2010 Nov 10. PMID 21074258
- [Background] Yusuf S, Reddy S, Ounpuu S, Anand S. Global burden of cardiovascular diseases: part I: general considerations, the epidemiologic transition, risk factors, and impact of urbanization. Circulation. 2001 Nov 27;104(22):2746-53. doi: 10.1161/hc4601.099487. PMID 11723030
- [Background] Lee DS, Chiu M, Manuel DG, Tu K, Wang X, Austin PC, Mattern MY, Mitiku TF, Svenson LW, Putnam W, Flanagan WM, Tu JV; Canadian Cardiovascular Outcomes Research Team. Trends in risk factors for cardiovascular disease in Canada: temporal, socio-demographic and geographic factors. CMAJ. 2009 Aug 4;181(3-4):E55-66. doi: 10.1503/cmaj.081629. Epub 2009 Jul 20. PMID 19620271
- [Background] Yusuf S, Islam S, Chow CK, Rangarajan S, Dagenais G, Diaz R, Gupta R, Kelishadi R, Iqbal R, Avezum A, Kruger A, Kutty R, Lanas F, Lisheng L, Wei L, Lopez-Jaramillo P, Oguz A, Rahman O, Swidan H, Yusoff K, Zatonski W, Rosengren A, Teo KK; Prospective Urban Rural Epidemiology (PURE) Study Investigators. Use of secondary prevention drugs for cardiovascular disease in the community in high-income, middle-income, and low-income countries (the PURE Study): a prospective epidemiological survey. Lancet. 2011 Oct 1;378(9798):1231-43. doi: 10.1016/S0140-6736(11)61215-4. Epub 2011 Aug 26. PMID 21872920
- [Background] Tu JV, Donovan LR, Lee DS, Wang JT, Austin PC, Alter DA, Ko DT. Effectiveness of public report cards for improving the quality of cardiac care: the EFFECT study: a randomized trial. JAMA. 2009 Dec 2;302(21):2330-7. doi: 10.1001/jama.2009.1731. Epub 2009 Nov 18. PMID 19923205
- [Background] Ahmad M, Schwalm JD, Velianou JL, Natarajan MK. Impact of routine in-hospital assessment of low-density lipoprotein levels and standardized orders on statin therapy in patients undergoing percutaneous coronary interventions. J Invasive Cardiol. 2005 Oct;17(10):518-20. PMID 16204743
- [Background] Newby LK, LaPointe NM, Chen AY, Kramer JM, Hammill BG, DeLong ER, Muhlbaier LH, Califf RM. Long-term adherence to evidence-based secondary prevention therapies in coronary artery disease. Circulation. 2006 Jan 17;113(2):203-12. doi: 10.1161/CIRCULATIONAHA.105.505636. Epub 2006 Jan 9. PMID 16401776
- [Background] Hudson M, Richard H, Pilote L. Parabolas of medication use and discontinuation after myocardial infarction--are we closing the treatment gap? Pharmacoepidemiol Drug Saf. 2007 Jul;16(7):773-85. doi: 10.1002/pds.1414. PMID 17486661
- [Background] Shah ND, Dunlay SM, Ting HH, Montori VM, Thomas RJ, Wagie AE, Roger VL. Long-term medication adherence after myocardial infarction: experience of a community. Am J Med. 2009 Oct;122(10):961.e7-13. doi: 10.1016/j.amjmed.2008.12.021. Epub 2009 Jun 26. PMID 19560749
- [Background] Rasmussen JN, Chong A, Alter DA. Relationship between adherence to evidence-based pharmacotherapy and long-term mortality after acute myocardial infarction. JAMA. 2007 Jan 10;297(2):177-86. doi: 10.1001/jama.297.2.177. PMID 17213401
- [Background] Rublee DA, Chen SY, Mardekian J, Wu N, Rao P, Boulanger L. Evaluation of cardiovascular morbidity associated with adherence to atorvastatin therapy. Am J Ther. 2012 Jan;19(1):24-32. doi: 10.1097/MJT.0b013e3181ee707e. PMID 20838204
- [Background] Shalev V, Chodick G, Silber H, Kokia E, Jan J, Heymann AD. Continuation of statin treatment and all-cause mortality: a population-based cohort study. Arch Intern Med. 2009 Feb 9;169(3):260-8. doi: 10.1001/archinternmed.2008.552. PMID 19204217
- [Background] Rodriguez LA, Cea-Soriano L, Martin-Merino E, Johansson S. Discontinuation of low dose aspirin and risk of myocardial infarction: case-control study in UK primary care. BMJ. 2011 Jul 19;343:d4094. doi: 10.1136/bmj.d4094. PMID 21771831